CLINICAL TRIAL: NCT03913637
Title: Influence of Strategy Training on Disability for Older Adults With Mild Cognitive Impairment
Brief Title: Facilitating Optimal Routines in Aging
Acronym: ForAging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Juleen Rodakowski, Associate Professor and Chair, Department of Occupational Therapy, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19120012; R01AG056351 (NIH)
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognition; Disability; Non-pharmacological Intervention; Behavioral Intervention; Amyloid deposition
MeSH Terms: conditions — Cognitive Dysfunction; Amyloidosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strategy Training (Experimental): In addition to receiving everything in Enhanced Usual Care, participants will engage in 10 sessions over 5 weeks with a trained research interventionist. Participants will describe activities they do, no longer do, or have never done using the cards from the Activity Card Sort as a guide. The therapist will ask the participants to use this information to identify and prioritize activity-based goals to address in the remaining sessions. These sessions will take place in a location of the participant's choice and will last approximately 1 hour.
  Interventions: Behavioral: Strategy Training
- Enhanced Usual Care (Active Comparator): Enhanced usual care will allow older adults to interact with services and support. All mental health treatment (e.g., medications that you may be taking) and psychotherapy (e.g. counseling or social services) will be documented and monitored. Furthermore, all participants assigned to Enhanced Usual Care will receive the same assessments as other participants. The close monitoring will track potential changes in symptoms (e.g., depressive symptoms), and participants will be referred to services as appropriate.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Strategy Training — Occupational therapists deliver Strategy Training to older adults virtually. Strategy training optimizes engagement in meaningful daily activities through generating self-selected goals, monitoring daily activities, scheduling activities, and problem-solving solutions to barriers experienced when engaging in activities.
  Arms: Strategy Training
Other: Enhanced Usual Care — In this comparison condition, usual care will be enhanced by connecting older adults with MCI to resources available to meet their needs, and notify appropriate physicians when required. Enhanced Usual Care provides a usual care comparison while providing the participants with close monitoring of changes in symptoms.
  Arms: Enhanced Usual Care

SUMMARY:
Loss of cognitive abilities leading to Alzheimer's disease is progressive and destructive, leaving older adults disabled and unable to recall their past. The number of older adults with Alzheimer's disease is expected to triple by the year 2050, yet little research examines amyloid beta deposition, executive function, and progression of disability. This study will test the influence of a novel and promising non-pharmacological intervention, Strategy Training, on the progression of disability in a sample of 150 older adults with Mild Cognitive Impairment who have the option to complete a Positron Emission Tomography (PET) Imaging with Pittsburgh Compound B (PiB).

DETAILED DESCRIPTION:
This trial will test the effect of Strategy Training compared to Enhanced Usual Care on change in disability among older adults with Mild Cognitive Impairment (MCI) and assess the extent to which Central Nervous System amyloid-beta deposition and neurocognitive function modify the relationship between Strategy Training and Enhanced Usual Care on change in disability. Assessments will be obtained at Baseline, 8 week short assessment, 6 and 12 months post intervention. Interventions, such as Strategy Training, focused on slowing emergence of disability despite underlying pathology may keep older adults as engaged in meaningful daily activities for as long as possible. This project tests a novel and promising non-pharmacological intervention and will inform our understanding of important effect modifiers- amyloid beta deposition and executive function- on change in performance of cognitively challenging daily activities. Enhancing our understanding of amyloid beta deposition, executive function, disability, and a promising non-pharmacological intervention could support aging for millions of older adults who, in the near future, will experience disability related to MCI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment
* Acknowledge difficulty with a daily activity
* Community dwelling

Exclusion Criteria:

* Pregnant
* Central Nervous System disorder (other than MCI)
* Substance disorder in past 5 years
* Lifetime history of bipolar disorder, schizophrenia, or deemed unsafe to proceed in the study (e.g., untreated Major Depressive Disorder)
* Severe medical condition that limits engagement in daily activities

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Change in disability | Baseline to Month 12
  Disability will be measured with the Performance Assessment of Self-Care Skills (PASS) through standardized, criterion-referenced performance assessment of cognitively challenging daily activities (i.e., shopping, bill paying, checkbook balancing, bill mailing, telephone use, medication management, critical information retrieval, and small device repair). A trained and blinded assessor will provide instruction and then observe participants performing each task. If the participant demonstrates difficulty, the assessor provides cues to assist. Assessors will rate disability based on the number of cues needed by the participants to complete the tasks. A higher score indicates more cues provided to complete the tasks or disability. The number of cues required for each task will be combined for a total number of cues provided on all 8 tasks. The outcome will be reported with a mean number of cues provided (range 0-300).

CONTACTS AND LOCATIONS:
Overall Officials: Juleen Rodakowski, OTD,MS,OTR/L, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will be included on The Global Alzheimer's Association Interactive Network (GAAIN). It is an operational online integrated research platform, which links scientists, shared data, and sophisticated analysis tools. Investigators can address scientific questions of unprecedented complexity by accessing massive shared data sets and can share their own data by joining our global network of Alzheimer's disease study centers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal.
URL: http://www.gaain.org